CLINICAL TRIAL: NCT02299206
Title: Randomized, Double-Blind, Parallel Group, Non-Inferiority Clinical Trial of CeraVe Baby Diaper Rash Cream Compared to Desitin Maximum Strength Original Paste for Management of Diaper Dermatitis in Infants
Brief Title: CeraVe Cream Compared to Desitin Paste for Treating Diaper Dermatitis in Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator and sponsor agreed to termination.
Sponsor: Northwestern University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Department of Dermatology, Professor of Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASP05012014
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CeraVe Baby Diaper Rash Cream (Experimental): Healthy 3-18 months old infants with mild to moderate diaper dermatitis.
  Interventions: Drug: CeraVe Baby Diaper Rash Cream
- Desitin Maximum Strength Original Paste (Experimental): Healthy 3-18 months old infants with mild to moderate diaper dermatitis.
  Interventions: Drug: Desitin Maximum Strength Original Paste

INTERVENTIONS:
Drug: CeraVe Baby Diaper Rash Cream — Parents/caregivers of subjects will administer CeraVe Baby Diaper Rash Cream (ingredients: Zinc oxide 10mg in 1g (1%) and dimethicone 10mg in 1g) with each diaper change throughout the course of the study period. The product can be applied liberally as needed. Diapers and skin cleansing interventions will stay constant throughout the treatment period.
  Other Names: CeraVe BDRC NDC Code: 0187-2221
  Arms: CeraVe Baby Diaper Rash Cream
Drug: Desitin Maximum Strength Original Paste — Parents/caregivers of subjects will administer Desitin Maximum Strength Original Paste (ingredients: Zinc Oxide 40%) with each diaper change throughout the course of the study period. The product can be applied liberally as needed. Diapers and skin cleansing interventions will stay constant throughout the treatment period.
  Other Names: Desitin MSOP NDC Code: 58232-0721
  Arms: Desitin Maximum Strength Original Paste

SUMMARY:
This is a single-center, 1:1 randomized, double-blind, parallel-group, non-inferiority controlled trial to demonstrate non-inferiority of CeraVe Baby Diaper Rash Cream compared to Desitin Maximum Strength Original Paste when administered to children with diaper dermatitis who are between 3 months to 18 months of age. Parents/caregivers of subjects in both groups will administer the product with each diaper change throughout the course of the study period. Product can be applied liberally as needed. Diapers and skin cleansing interventions will stay constant throughout the treatment period. Subjects will be assessed by the study doctor, parent/caregiver will be asked about any adverse effects. Parent/caregivers will also be asked to complete a daily diary that asks about changes in their baby's diaper dermatitis, a Visual Analogue Scale severity assessment of their baby's diaper dermatitis, and observations related to product use and the baby's comfort level. Parents/caregivers will also be given a questionnaire rating the use of the study products.

DETAILED DESCRIPTION:
Visit 1 - Screening and Baseline Visit (Day 0) Subjects will be evaluated for study eligibility using inclusion and exclusion criteria. The study doctor will assess diaper dermatitis for inclusion and exclusion criteria and to verify mild to moderate severity. Once study eligibility has been confirmed, parental/guardian consent will be obtained. No washout period is necessary for this study.

Location of clinically apparent involved area will be shaded by hand onto diagram by the research personnel. Study products will be dispensed to parent/caregiver, along with instructions for administration. Parent/caregivers will also be asked to complete a daily diary that asks about changes in their baby's diaper dermatitis, a Visual Analogue Scale severity assessment of their baby's diaper dermatitis, and observations related to product use and the baby's comfort level. Parents/caregivers will be asked to complete the daily diary for each day of the study.

Visit 2 (Day 7) Subjects will again be assessed by the study doctor. Parent/caregiver will be asked about any adverse effects in last 7 days.

Visit 3 - End of study (Day 14) Subjects will again be assessed by the study doctor. Daily diaries and product will be collected at this time. Parent/caregiver will be asked about any adverse effects in last 7 days. Parents/caregivers will also be given a questionnaire rating the use of the study products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (except for diaper dermatitis) between 3 and 18 months of age
* Wearing diapers 24 hours per day
* Clinical irritant diaper dermatitis
* Received a Diaper Dermatitis severity score of 1.0 to 2.0 by investigator at screening visit (mild-moderate severity)
* Parent/caregiver will not change type or brand of diaper during the study, although the diaper type will be recorded
* No alteration of current product usage for creams, lotions, ointments, powders, soap, laundry detergents, and fabric softeners
* A parent or guardian of minors must sign the approved Institutional Review Board consent form prior to the conduct of any study-related procedures

Exclusion Criteria:

* Illness within past 4 days before study enrollment or any medical condition that may affect risk of study participation
* Does not wear diapers 24 hours per day or currently being toilet trained
* Active diagnosis or history of dermatological conditions other than diaper rash that may affect study
* Concomitant use of medications that may affect study (e.g., antifungal, topical steroid, or topical calcineurin inhibitor)
* Previous allergic reaction or known sensitivity to ingredients in study agents

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Department of Der,matology, Feinberg School of Medicine, Northwestern University
Locations (3):
- United States (3):
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University Department of Dermatology, Chicago, Illinois
  - Lurie Children's Hospital Outpatient Clinic at Lincoln Park, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arms are combined for overall number of participants. Due to the low number of subjects, data will not be analyzed and the arm assignment for the subjects was not determined.
Groups:
- CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina: Healthy 3-18 months old infants with mild to moderate diaper dermatitis.
  CeraVe Baby Diaper Rash Cream: Parents/caregivers of subjects will administer CeraVe Baby Diaper Rash Cream (ingredients: Zinc oxide 10mg in 1g (1%) and dimethicone 10mg in 1g) or Desitin Maximum Strength Original Paste (ingredients: Zinc Oxide 40%) with each diaper change throughout the course of the study period. The product can be applied liberally as needed. Diapers and skin cleansing interventions will stay constant throughout the treatment period.
Period: Overall Study
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Started | 4
Completed | 2
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Arms are combined for overall number of baseline participants. Due to the low number of subjects, data will not be analyzed and the arm assignment for the subjects was not determined.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: months] | 11.5 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for the Physician Assessment Diaper Dermatitis Scores to Day 14 for Each Treatment Group.
Description: For each visit the study doctor will assess the diaper dermatitis severity with a Diaper Dermatitis Severity Score tool. In Addition, location of clinically apparent involved area will be shaded by hand onto diagram by the research personnel. Scores will be compared.
Time Frame: 14 days
Population: Study was terminated prior to analysis due to low enrollment.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Physician Assessment Diaper Dermatitis Scores to Day 7
Description: as for outcome 1
Time Frame: 7 days
Population: Study was terminated prior to analysis due to low enrollment.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 0

3. Secondary Outcome: Parents/Caregivers Daily Scores Through Duration of the Study Period
Description: Parent/caregivers will be asked to complete a daily diary that asks about changes in their baby's diaper dermatitis, a Visual Analogue Scale severity assessment of their baby's diaper dermatitis, and observations related to product use and the baby's comfort level
Time Frame: 14 days
Population: Study was terminated prior to analysis due to low enrollment.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 0

4. Secondary Outcome: Assessment of Tolerability by the Infant
Description: Parent/caregivers will be asked to complete a daily diary that asks about changes in their baby's diaper dermatitis, a VAS severity assessment of their baby's diaper dermatitis, and observations related to product use and the baby's comfort level
Time Frame: 14 days
Population: Study was terminated prior to analysis due to low enrollment.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 0

5. Secondary Outcome: Parent/Caregiver Rating of Satisfaction With Use of the Product
Description: Parents/caregivers will be given a questionnaire rating the use of the study products.
Time Frame: 14 days
Population: Study was terminated prior to analysis due to low enrollment.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina: Healthy 3-18 months old infants with mild to moderate diaper dermatitis.
  CeraVe Baby Diaper Rash Cream: Parents/caregivers of subjects will administer CeraVe Baby Diaper Rash Cream (ingredients: Zinc oxide 10mg in 1g (1%) and dimethicone 10mg in 1g) or Desitin Maximum Strength Original Paste (ingredients: Zinc Oxide 40%) with each diaper change throughout the course of the study period. The product can be applied liberally as needed. Diapers and skin cleansing interventions will stay constant throughout the treatment period.
  Arms are combined for reporting of adverse events. Due to the low number of subjects, data will not be analyzed and the arm assignment for the subjects was not determined.
Arm/Group | CeraVe Baby Diaper Rash Cream/Desitin Maximum Strength Origina
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes